CLINICAL TRIAL: NCT01278420
Title: AMO's Tecnis™ Multifocal Intraocular Lenses (Tecnis MF), Alcon's ReStor Multifocal IOL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovative Medical (Industry)
Responsible Party: William Trattler, The Center for Excellence in Eye Care
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMF vs Restor MF 3D
Record Dates: First submitted 2010-08-27; First posted 2011-01-17 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Cataract
Keywords: Visual outcomes with bilateral implantation of Tecnis MF and ReSTOR IOLs Six months post cataract surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tecnis MF (Other)
  Interventions: Device: Tecnis MF
- ReSTOR (Other)
  Interventions: Device: ReSTOR

INTERVENTIONS:
Device: Tecnis MF — 30 subjects will be implanted with the Tecnis MF
  Arms: Tecnis MF
Device: ReSTOR — 30 subjects will be implanted with ReSTOR
  Arms: ReSTOR

SUMMARY:
The purpose of this study is to compare the visual outcomes with bilateral implantation of Tecnis MF and ReSTOR IOLs Six months post cataract surgery.

DETAILED DESCRIPTION:
The purpose of this study is to compare the visual outcomes with bilateral implantation of Tecnis MF and ReSTOR IOLs Six months post cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Bilateral condition (cataracts or Presbyopia) for which phacoemulsification and posterior IOL implantation has been planned for both eyes
* Visual potential of 20/25 or better in each eye after cataract removal and IOL implantation
* Clear intraocular media other than cataract
* Normal OCT of the macula
* No evidence of Keratoconus or significant irregular astigmatism on Preoperative topography
* No evidence of Epithelial Basement Membrane Dystrophy on Slit lamp Exam
* Availability, willingness, and sufficient cognitive awareness to comply with examination procedures

Exclusion Criteria:

* Use of systemic or ocular medications that may affect vision
* Uncontrolled systemic or ocular disease
* History of ocular trauma
* History of intraocular, extraocular Muscle, or corneal surgery (including laser vision correction)
* Amblyopia or strabismus
* Known pathology that may affect visual acuity; particularly retinal changes that affect vision (macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, etc.)
* Diagnosed degenerative visual disorders (e.g. macular degeneration, or other retinal disorders) that are predicted to cause future acuity losses to a level of 20/25 or worse
* Subjects who may be expected to require retinal laser treatment or other surgical intervention (i.e patients with diabetic retinopathy)
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome)
* Contact lens usage within 2 months for PMMA contacts lenses, 2 weeks for gas permeable lenses or 3 days for extended-wear and daily-wear soft contact lenses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Refraction | 1 year
Distance Visual Acuities | 1 year
Near Visual Acuities | 1 year
Intermediate Acuities | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: William Trattler, MD, Principal Investigator — The Center for Excellence in Eye Care; Mitch Jackson, MD, Principal Investigator — Jackson Eye; Larry Katzen, MD, Principal Investigator — Katzen Eye Care & Laser Center; Kevin Waltz, MD, Principal Investigator — Eye Surgeons of Indiana; Shamik Bafna, MD, Principal Investigator — Clevland Eye Clinic
Locations (6):
- United States (6):
  - Sansum- Santa Barbara medical foundation Clinic, Santa Barbara, California
  - Katzen Eye Care & Laser Center, Boynton Beach, Florida
  - The Center for Excellence in Eye Care, Miami, Florida
  - Jackson Eye, SC, Lake Villa, Illinois
  - Eye Surgeons of Indiana, Indianapolis, Indiana
  - Cleveland Eye Clinic, Breckville, Ohio